CLINICAL TRIAL: NCT05878496
Title: Short Term Outcome of Pediatric Fracture of Neck Femur Fixation by Plate and Screws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Hussien Ahmed, short term outcome of pediatric fracture of neck femur fixation by plate and screws, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-22MS
Record Dates: First submitted 2023-05-07; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Fracture of Pediatric Neck Femur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: fixation by plate and screws — reduction and fixation of pediatric fracture neck femur by plate and screws

SUMMARY:
the incidence of femoral neck fracture in children ranges between 0.3 and 0.5 of all childhood fractures per year. the incidence is maximum at the ranges of 11 and 12 years with a male preponderance ranging from 1.3 to 1.7:1. in contrast to osteoprotic proximal femur fractures in the eldery. although rarely seen in children fracture neck of femur has aconsiderable risk of complications such as avascular necrosisos femoral head, coxa vara, non union, delayed union, premature physeal arrest and infection. in infants and toddlrs below age of 2 years, closed reduction and fixation with smooth 1.8 or 2 mm K wires may be carried out, in children there are many methods of fixation, cannulated 4,4.5 screws, plates,dynamic hip screw.

DETAILED DESCRIPTION:
the incidence of femoral neck fracture in children ranges between 0.3 and 0.5 of all childhood fractures per year. the incidence is maximum at the ranges of 11 and 12 years with a male preponderance ranging from 1.3 to 1.7:1. in contrast to osteoprotic proximal femur fractures in the eldery. although rarely seen in children fracture neck of femur has aconsiderable risk of complications such as avascular necrosisos femoral head, coxa vara, non union, delayed union, premature physeal arrest and infection. in infants and toddlrs below age of 2 years, closed reduction and fixation with smooth 1.8 or 2 mm K wires may be carried out, in children there are many methods of fixation, cannulated 4,4.5 screws, plates,dynamic hip screw.

ELIGIBILITY:
Inclusion Criteria:

* children between 2 and 16 years having fracture of neck femur

Exclusion Criteria:

* patients more than 16 years, cases with open fractures, preexisting deformity, other pelvic or ipsilateral femoral injuries

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
avascular necrosis by degree of bone necrosis in head and neck femur | 6 months
  osteonecrosis and death of bone tissue of head and neck femur

SECONDARY OUTCOMES:
coxa vara degree by angle of shaft and head femur | 6 months
  angle between the head and the shaft femur is reduced to less than 120 degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Patterson JT, Tangtiphaiboontana J, Pandya NK. Management of Pediatric Femoral Neck Fracture. J Am Acad Orthop Surg. 2018 Jun 15;26(12):411-419. doi: 10.5435/JAAOS-D-16-00362. PMID 29781820
- [Background] RATLIFF AH. Fractures of the neck of the femur in children. J Bone Joint Surg Br. 1962 Aug;44-B:528-42. doi: 10.1302/0301-620X.44B3.528. No abstract available. PMID 14038616
- [Background] Mirdad T. Fractures of the neck of femur in children: an experience at the Aseer Central Hospital, Abha, Saudi Arabia. Injury. 2002 Nov;33(9):823-7. doi: 10.1016/s0020-1383(02)00013-x. PMID 12379394
- [Background] Azouz EM, Karamitsos C, Reed MH, Baker L, Kozlowski K, Hoeffel JC. Types and complications of femoral neck fractures in children. Pediatr Radiol. 1993;23(6):415-20. doi: 10.1007/BF02012436. PMID 8255640